CLINICAL TRIAL: NCT01269762
Title: Pharmacokinetic and Drug Interaction Study of Red Yeast Rice Capsules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201001003M
Record Dates: First submitted 2010-12-21; First posted 2011-01-04 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Volunteer
Keywords: Red yeast rice; Lovastatin; Drug-drug interaction; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LipoCol Forte (Experimental): Subject will receive single dose of one, two and four 600 milligram (mg) red yeast rice capsules (LipoCol Forte)and multiple dose of 600 mg red yeast rice Capsules (LipoCol Forte)twice daily for 4.5 days.
  Interventions: Drug: LipoCol Forte

INTERVENTIONS:
Drug: LipoCol Forte — Single dose of one, two and four 600 mg red yeast rice capsules (LipoCol Forte) Multiple dose of 600 mg red yeast rice Capsules (LipoCol Forte)twice daily for 4.5 days

SUMMARY:
Red yeast rice capsule (LipoCol Forte)is a nature product that has been demonstrated a significant cholesterol lowering effect which might be caused by addictive and/or synergistic effects of lovastatin (monacolin K) with other monacolins and substances in capsules. The usual dose of red yeast rice capsule(LipoCol Forte)for hypercholesterolemia is one capsule twice/day.

However, the pharmacokinetic profile of red yeast rice capsule (LipoCol Forte)is still unknown.

The objective of the study is to evaluate the pharmacokinetic profile of red yeast rice capsule (LipoCol Forte) after administering single and multiple dose to healthy subjects.

DETAILED DESCRIPTION:
This study will divide into two groups, single and multiple doses groups. In single dose group, the subjects will receive one, two and four red yeast rice capsules under fed state in period one to three, respectively. In multiple doses group, the subjects will receive red yeast rice capsules under fed state twice daily for 4.5 days. There is a minimum of a 5-days washout period before crossover of treatments.

In single dose treatment, the blood samples will be drawn prior to the dosing, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours after the dosing.

In multiple doses treatment, the blood samples will be drawn prior to the 1st dosing, prior to the 7th dosing, prior to the 8th dosing, prior to the 9th dosing, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours after the 9th dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at the age of 20-40 years old and in good health on the basis of medical history, physical examination, electrocardiogram, chest X-ray, and routine laboratory evaluations.
2. Vital signs (after 3 minutes resting in a upright position) which are within the following ranges:

   Ear body temperature between 35.0-37.5 degree celsius (°C). Systolic blood pressure, 90-140 millimeters of mercury (mm Hg). Diastolic blood pressure, 50-90 millimeters of mercury (mm Hg). Pulse rate, 50-90 beats per minute (bpm). Fasting blood glucose, < 110 milligrams per deciliter (mg/dL).
3. Body weight must be above 50 kilograms (kg) and within -20 to +20% of ideal body weight.
4. Able to sign informed consent prior to study.

Exclusion Criteria:

1. Use of any prescription medication within 14 days prior to dosing.
2. Use of over-the-counter medications or vitamins within 14 days prior to dosing.
3. Participation in any clinical investigation within 3 months prior to dosing or longer as required by local regulation.
4. Donation or loss of more than 500 milliliter (mL) blood within 3 months prior to dosing.
5. Significant illness within 2 weeks prior to dosing.
6. Presence of cardiovascular diseases.
7. Presence of gastrointestinal diseases.
8. Presence of asthma or lung diseases.
9. Presence of liver disease or liver injury.
10. Presence of impaired renal function.
11. Presence of neurological diseases.
12. Presence of psychiatrical diseases.
13. Subject is known for Human Immunodeficiency Virus (HIV) infected.
14. A known hypersensitivity to lovastatin or its analogs.
15. History of drug or alcohol abuse within 12 months prior to dosing.
16. Permanent confinement to an institution.
17. Individuals are judged by the investigator or co-investigator to be undesirable as subjects for other reasons.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The maximum tolerate dosage | 5 weeks
  The maxium tolerate dosage

SECONDARY OUTCOMES:
Evaluation of the pharmacokinetic parameters of LipoCol Forte in healthy subjects | 5 weeks
  Evaluation of pharmacokinetic parameters of LipoCol Forte in healthy subjects after single and multiple doses
The incidence rate of adverse event | 5 weeks
  The incidence rate of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jyh-Chin, M.D. Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan